CLINICAL TRIAL: NCT05323422
Title: EFFECT OF LOW DOSE INTRAVENOUS KETAMINE ON POSTOPERATIVE COGNITIVE FUNCTIONS
Brief Title: EFFECT OF LOW DOSE INTRAVENOUS KETAMINE GIVEN BEFORE INDUCTION ON POSTOPERATIVE COGNITIVE FUNCTIONS IN PATIENTS WITH COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, medical doctor, Kocaeli Derince Education and Research Hospital
Other Study IDs: 2021-514-214-38
Record Dates: First submitted 2022-04-11; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pandemic
Keywords: Covid-19, Ketamine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: COVID-19 positive and pre-induction low-dose intravenous ketamine (0.5 mg/kg) will administering
  Interventions: Procedure: intravenous Ketamine induction
- Group 2: COVID-19 positive and without intravenous ketamine (0.5 mg/kg)
- Group -3: COVID-19 negative and pre-induction low-dose intravenous ketamine (0.5 mg/kg) will administering
  Interventions: Procedure: intravenous Ketamine induction
- Group4: COVID-19 negative and without intravenous ketamine (0.5 mg/kg)

INTERVENTIONS:
Procedure: intravenous Ketamine induction — preoperatively ketamine wll administer in group 1-3
  Groups: Group -3; Group 1

SUMMARY:
Postoperative psychomotor dysfunction is called postoperative cognitive dysfunction, and the incidence of postoperative complications is high, especially in elderly patients undergoing major surgery. This complication; It can be attributed to the anesthetic agents used, their doses, and the duration of the surgery. Although SARS-CoV-2 virus causes an infection called Covid-19 that mainly affects the respiratory tract, data have been obtained that it can enter the nasal mucosa, reach the central nervous system via olfactory fibers or hematogenous way, and infect endothelial cells and neurons. The immune system is activated due to endothelial cell damage, vascular permeability increases, and the risk of thrombosis occurs. Cerebral hypoperfusion promotes Lewy body development, especially by increasing amyloid plaque formation and inducing serine phosphorylation. The formation of these plaques, which are responsible for the development of Alzheimer's and Dementia, suggests that Covid-19 may have long-term neurological complications. In our study, we included patients who were scheduled for cholecystectomy, who had and did not have covid-19 infection. Covid-19 infection (Group 1), no previous (Group 2), COVID-19 and pre-induction low-dose intravenous ketamine (0.5 mg/kg) administered (Group 3), non-covid-19 and pre-induction low-dose intravenous ketamine We aimed to evaluate and compare postoperative cognitive functions in patients (Group 4) administered (0.5 mg/kg). Ketamine is a sedative, hypnotic and analgesic agent and has an effective role in balanced anesthesia. In addition, its use reduces the need for the use of other anesthetic agents. The use of ketamine in normal doses causes a decrease in brain and cognitive functions; The use of sub-anesthetic doses before induction has positive effects on recovery and cognitive functions. Depth of anesthesia with bispectral index continuously before and throughout the operation; The lowest and highest values were recorded by regional cerebral oximetry (rSO2) measurement. Cognitive tests were performed 1 day before the operation, at the 12th hour and 30 days after the operation. MMT (mini mental test), Verbal Fluency Test (verbal fluency test), Clock Drawing Test (clock drawing test) Aldrete recovery scores were evaluated at the 2nd and 5th minutes after extubation. The study included 160 patients, 35-55 young and middle-aged, ASA I and II. Patients who underwent emergency surgery, had malignancy, and had a known chronic disease were excluded from the study.

DETAILED DESCRIPTION:
Postoperative psychomotor dysfunction is called postoperative cognitive dysfunction, and the incidence of postoperative complications is high, especially in elderly patients undergoing major surgery. This complication; It can be attributed to the anesthetic agents used, their doses, and the duration of the surgery. Although SARS-CoV-2 virus causes an infection called Covid-19 that mainly affects the respiratory tract, data have been obtained that it can enter the nasal mucosa, reach the central nervous system via olfactory fibers or hematogenous way, and infect endothelial cells and neurons. The immune system is activated due to endothelial cell damage, vascular permeability increases, and the risk of thrombosis occurs. Cerebral hypoperfusion promotes Lewy body development, especially by increasing amyloid plaque formation and inducing serine phosphorylation. The formation of these plaques, which are responsible for the development of Alzheimer's and Dementia, suggests that Covid-19 may have long-term neurological complications. In our study, we included patients who were scheduled for cholecystectomy, who had and did not have covid-19 infection. Covid-19 infection (Group 1), no previous (Group 2), COVID-19 and pre-induction low-dose intravenous ketamine (0.5 mg/kg) administered (Group 3), non-covid-19 and pre-induction low-dose intravenous ketamine We aimed to evaluate and compare postoperative cognitive functions in patients (Group 4) administered (0.5 mg/kg). Ketamine is a sedative, hypnotic and analgesic agent and has an effective role in balanced anesthesia. In addition, its use reduces the need for the use of other anesthetic agents. The use of ketamine in normal doses causes a decrease in brain and cognitive functions; The use of sub-anesthetic doses before induction has positive effects on recovery and cognitive functions. Depth of anesthesia with bispectral index continuously before and throughout the operation; The lowest and highest values were recorded by regional cerebral oximetry (rSO2) measurement. Cognitive tests were performed 1 day before the operation, at the 12th hour and 30 days after the operation. MMT (mini mental test), Verbal Fluency Test (verbal fluency test), Clock Drawing Test (clock drawing test) Aldrete recovery scores were evaluated at the 2nd and 5th minutes after extubation. The study included 160 patients, 35-55 young and middle-aged, ASA I and II. Patients who underwent emergency surgery, had malignancy, and had a known chronic disease were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35-55 years ASA 1, 2 group Patients scheduled for cholecystectomy

Exclusion criteria:

Patient's refusal to participate in the study Those with malignancy Patients scheduled for emergency surgery

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with and without covid 19
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-04-12 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of cognitive function | 6 months
  Cognitive functions will be evaluated after induction with ketamine in patients with and without covid 19

IPD SHARING:
Plan to Share IPD: No